CLINICAL TRIAL: NCT02704416
Title: Ablation in Brugada Syndrome for Prevention of VF - A Randomized, Multi-center Study of Epicardial Ablation in Brugada Syndrome Patients to Prevent Arrhythmia Recurrence
Brief Title: Ablation in Brugada Syndrome for the Prevention of VF
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Rim Electrophysiology Research Institute (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Koonlawee Nademanee, MD, Principal Investigator, Pacific Rim Electrophysiology Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PacificRERI
Record Dates: First submitted 2016-02-18; First posted 2016-03-10 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Brugada Syndrome
Keywords: Ventricular arrhythmias; aborted cardiac arrest; cardiac death
MeSH Terms: conditions — Brugada Syndrome; Death | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control arm (No Intervention): Control arm - continued implanted cardioverter defibrillator therapy
- Intervention Arm (Active Comparator): ablation of areas of fragmented signal in the right ventricular outflow tract plus continued implanted cardioverter defibrillator therapy
  Interventions: Procedure: Catheter Ablation
- Single Cross Over Arm (Other): these patients were initially assigned to the control arm of the study. When these patients met the primary outcome of the study it is allowed for these patients to be included in the intervention arm and/or to start quinidine
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — catheter ablation of fragmented signal in the right ventricular outflow tract
  Arms: Intervention Arm; Single Cross Over Arm

SUMMARY:
This trial aims to develop evidence based curative treatment with optimal net benefit for patients with Brugada syndrome.

DETAILED DESCRIPTION:
This trial aims to develop evidence based curative treatment with optimal net benefit for patients with Brugada syndrome. Since a recent non-randomized pilot study and scarce case reports documented potential clinical benefit of epicardial ablation of fragmented electrograms in the region of the right ventricular outflow tract, patients in this trial will be randomized to continued implanted cardioverter defibrillator therapy (control arm) or ablation of areas of fragmented electrograms in the right ventricular outflow tract plus continued implanted cardioverter defibrillator therapy (intervention arm). A projected 92 patients in each group will be studied.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Brugada syndrome is based on 2013 HRS/EHRA/APHRS Consensus document criteria
* Diagnosed symptomatic BrS with an implanted ICD within the last 5 years
* Diagnosed symptomatic BrS with an implanted ICD longer than 5 years but has at least 1 appropriate shock within the last 5 years
* The patient is legally competent, willing and able to undergo the study and signed the informed consent
* The patient is willing and able to adhere to the follow-up visit protocol

Exclusion Criteria:

* A patient who does not meet inclusion criteria
* A patient who has had a previous epicardial ablation
* A patient who is pregnant (which would exclude an ablation procedure)
* A patient with a co-morbid condition that possesses undue risk of general anesthesia or epicardial ablation
* A patient who has a history of radiation therapy on the thorax

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07; Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Freedom of Ventricular Fibrillation/Tachycardia Recurrences | 3 year followup
  Survival from ventricular fibrillation of shocked ventricular arrhythmias causing ICD discharge

SECONDARY OUTCOMES:
Freedom without drug | 3 years
  Freedom of shocked ventricular arrhythmias without the use of anti-arrhythmic drugs during 3 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Koonlawee Nademanee, MD, Principal Investigator — Pacific Rim Electrophysiology Research Institute
Locations (6):
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands
- Thailand (5):
  - Bhumipol Adulyadej Hospital, Royal Thai Air Force, Bangkok
  - Chulalongkorn University, Bangkok
  - Pacific Rim Electrophysiology Research Institute Data Coordinating Center, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Chiang Mai University, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Medical journals, abstract submissions and results database

REFERENCES:
- [Background] Nademanee K, Raju H, de Noronha SV, Papadakis M, Robinson L, Rothery S, Makita N, Kowase S, Boonmee N, Vitayakritsirikul V, Ratanarapee S, Sharma S, van der Wal AC, Christiansen M, Tan HL, Wilde AA, Nogami A, Sheppard MN, Veerakul G, Behr ER. Fibrosis, Connexin-43, and Conduction Abnormalities in the Brugada Syndrome. J Am Coll Cardiol. 2015 Nov 3;66(18):1976-1986. doi: 10.1016/j.jacc.2015.08.862. PMID 26516000
- [Background] Nademanee K, Veerakul G, Chandanamattha P, Chaothawee L, Ariyachaipanich A, Jirasirirojanakorn K, Likittanasombat K, Bhuripanyo K, Ngarmukos T. Prevention of ventricular fibrillation episodes in Brugada syndrome by catheter ablation over the anterior right ventricular outflow tract epicardium. Circulation. 2011 Mar 29;123(12):1270-9. doi: 10.1161/CIRCULATIONAHA.110.972612. Epub 2011 Mar 14. PMID 21403098
- [Background] Ten Sande JN, Coronel R, Conrath CE, Driessen AH, de Groot JR, Tan HL, Nademanee K, Wilde AA, de Bakker JM, van Dessel PF. ST-Segment Elevation and Fractionated Electrograms in Brugada Syndrome Patients Arise From the Same Structurally Abnormal Subepicardial RVOT Area but Have a Different Mechanism. Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1382-92. doi: 10.1161/CIRCEP.115.003366. Epub 2015 Oct 19. PMID 26480928
- [Background] Wilde AA, Nademanee K. Epicardial Substrate Ablation in Brugada Syndrome: Time for a Randomized Trial! Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1306-8. doi: 10.1161/CIRCEP.115.003500. No abstract available. PMID 26671932